CLINICAL TRIAL: NCT06098859
Title: Comparison of the Effects of Thoracic Epidural Analgesia and Bilateral Erector Spinae Plane Block on Postoperative Pain and Respiratory Fonctions in Open Heart Surgeries''
Brief Title: Thoracic Epidural Analgesia and Bilateral Erector Spinae Plane Block on Postoperative Pain in Open Heart Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Engin Ertürk, Prof. Dr, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023/184
Record Dates: First submitted 2023-10-13; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Pain, Postoperative; Respiratory Complication
Keywords: Thoracic epidural analgesia; erector spinae plane block; heart surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Tea

STUDY DESIGN:
Intervention Model Description: The effects of thoracic epidural analgesia and erector spinae plane block on postoperative pain were compared with the control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants did not know which method was applied to them. Those who evaluated the research results did not know the groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Thoracic epidural analgesia (Active Comparator): Thoracic epidural analgesia have been started preoperatively and coninuoed until postoperative 48 hours
  Interventions: Procedure: Thoracic epidural analgesia
- Erector spinae plane block (Active Comparator): Erector spinae plane blockwas applied preoperatively
  Interventions: Procedure: Erector spinae plane block
- Intravenous opioid analgesia (No Intervention): Intravenous opioid analgesia was administered during the surgery

INTERVENTIONS:
Procedure: Thoracic epidural analgesia — Thoracic epidural analgesia was started preoperatively and rest posoperative 48 hours
  Arms: Thoracic epidural analgesia
Procedure: Erector spinae plane block — Erector spinae plane block was applied preoperatively using local anesthetic
  Arms: Erector spinae plane block

SUMMARY:
Postoperative pain negatively effects respiratory functions in open heart surgeries. The aim of the study is to compare the effects of thoracic epidural analgesia (TEA) and erector spinae plane block (ESPB) on postoperative pain and respiratory functions in patients undergoing open heart surgery with sternotomy

DETAILED DESCRIPTION:
Thoracic epidural catheter was inserted to patients in Group T at the T4-T5 vertebra level before induction of general anesthesia. And then local anesthetic infusion was started until postoperative 48. hours.

Bilateral erector spinae plan block was applied with total 40 ml of local anesthetic solution to patients in Group E at the T4-T5 vertebra level before induction of general anesthesia.

The control group was infused with 1 mcg/kg/min fentanyl during the surgery. In the postoperative period, 1 g paracetamol was infused 4 times a day.

All patients underwent general anesthesia with the same method and medications.

Tramadol/diclofenac was administered to patients with a pain score (NRS) above 4. NRS and tidal volumes (TV) of the patients were measured at 0, 2, 6, 12, 24, 36 and 48. hours after extubation. Postoperative mechanical ventilation durations, intensive care unit and hospital stays, additional analgesic needs and respiratory complications of the patients were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Has ASA II-IV score
* Having open heart surgery

Exclusion Criteria:

* Having a psychiatric illness
* Using analgesic medication due to chronic pain
* Uncooperative

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Postoperative 48 hours
  Patients were asked about their pain levels. Rating done with VRS (Verbal Rating Scale).
  Pain levels were evaluated between 0 and 10 points. 0: No pain (the best)….. 10: Unbearable pain (the worst)
Respiratory functions | Postoperative 48 hours
  Oxygen requirement:If more than 4 l/min oxygen support via face mask is required to maintain peripheral oxygen saturation (SpO2) above 90%, it is defined as oxygen requirement.
  Tachypnea:more than 20/min
  Fever: more than 37 C celcius
  Non invasive mechanical ventilation requirement:To patients whose breathing is impaired after extubation (who have tachypnea and have SpO2 less than 90% despite receiving oxygen support of more than 4 l/min oxygen support via face mask)

SECONDARY OUTCOMES:
Analgesic requirement. When the VRS was more than 4 points | Postoperative 48 hours
  diclofenac (75 mg), tramadol (50mg)
Intensive care and hospital stay | postoperative 30 days
  time for Intensive care and hospital (hours and days, respectively)

CONTACTS AND LOCATIONS:
Overall Officials: Engin Ertürk, Prof. Dr, Principal Investigator — Karadeniz Technical University, Medical Faculty, Anesthesiology and Intensive Care
Locations (1):
- Engin Ertürk, Ortahisar, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting12 months after publication
Access Criteria: analyst and investigators